CLINICAL TRIAL: NCT00287846
Title: Multicentric Phase I/II Study Evaluating the Efficacy and Toxicity of Imatinib in Adult Patients With Aggressive Fibromatosis That Cannot be Treated by Surgery or Curative Radiotherapy
Brief Title: Imatinib Mesylate in Treating Patients With Recurrent or Refractory Fibromatosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000441039; FRE-FNCLCC-SARCOME-05/0401; EU-20515
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Desmoid Tumor
Keywords: desmoid tumor
MeSH Terms: conditions — Desmoid Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Imatinib (Experimental): 400 to 800 mg/day for a maximal 12 months study duration.
  Interventions: Drug: imatinib mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
RATIONALE: Imatinib mesylate may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

PURPOSE: This phase I/II trial is studying the side effects of imatinib mesylate and to see how well it works in treating patients with recurrent or refractory aggressive fibromatosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the non-progression rate in patients with recurrent or refractory aggressive fibromatosis after 3 months of treatment with imatinib mesylate.

Secondary

* Determine the non-progression rate in patients after being treated with this drug for 12 months.
* Determine the toxic effects of this drug in these patients.
* Determine the tolerance to this drug in these patients.
* Determine the response rate in patients treated with this drug
* Determine progression free and overall survival of patients treated with this drug.
* Determine the quality of life of patients treated with this drug.
* Correlate clinical, biological, and genomic markers with response and long-term stable disease in patients treated with this drug.

OUTLINE: This is a multicenter study.

Patients receive oral imatinib mesylate once daily for up to 12 months in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed periodically.

PROJECTED ACCRUAL: A total of 39 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed aggressive fibromatosis (desmoid tumor)
* Relapse or disease progression despite surgery, chemotherapy, radiotherapy, or any other treatment
* Tumors must meet the following criteria:

  * Ineligible for complete surgical resection by carcinological exeresis OR surgery would cause severe mutilation
  * Cannot be treated with curative radiotherapy
* Measurable disease by RECIST criteria
* No prior malignancy

PATIENT CHARACTERISTICS:

* Not pregnant or nursing
* Fertile patients must use effective contraception during and for 6 months after completion of study treatment
* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm^3
* Bilirubin < 1.5 times upper limit of normal (ULN)
* SGOT and SGPT < 2.5 times ULN
* Creatinine ≤ 2.5 times normal
* No severe liver failure
* No chronic somatic or psychiatric illness that would preclude study compliance
* No known hypersensitivity to imatinib mesylate or one of its components
* No geographical, social, or psychological reason that would inhibit follow-up

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent immunomodulators*
* No concurrent hormonal treatments* if used for fibromatosis
* No concurrent cytotoxic drugs*
* No concurrent nonsteroidal anti-inflammatory drug* if used for fibromatosis

  * Allowed if used as an analgesic 3 months prior to disease progression
* No concurrent participation in another therapeutic investigational trial NOTE: *If disease progression has occurred during this treatment, then the treatment must have ended ≥ 1 month prior to study entry

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-09; Primary Completion 2006-02 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Non-progression rate | 3 months

SECONDARY OUTCOMES:
Non-progression rate | 12 months
Toxic effects | 12 months
Tolerance | 12 months
Response rate | 5 years
Progression-free survival | the time between the inclusion date and the progression date
Overall survival | the time between the inclusion date and the death whathever the cause
Quality of life | 5 years
Correlation of clinical, biological, and genomic markers with response and long-term stable disease | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Blay, MD, PhD, Study Chair — Hopital Edouard Herriot - Lyon
Locations (23):
- France (23):
  - Centre Paul Papin, Angers
  - Centre Hospitalier Regional de Besancon - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Regional Francois Baclesse, Caen
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Hopital Edouard Herriot - Lyon, Lyon
  - CHU de la Timone, Marseille
  - Centre Regional de Lutte Contre le Cancer - Centre Val d'Aurelle, Montpellier
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Curie Hopital, Paris
  - Hopital Tenon, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Hopitaux Universitaire de Strasbourg, Strasbourg
  - Hopital Foch, Suresnes
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau de Tours, Tours
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant data will not be shared at an individual level.

REFERENCES:
- [Result] Penel N, Le Cesne A, Bui BN, Perol D, Brain EG, Ray-Coquard I, Guillemet C, Chevreau C, Cupissol D, Chabaud S, Jimenez M, Duffaud F, Piperno-Neumann S, Mignot L, Blay JY. Imatinib for progressive and recurrent aggressive fibromatosis (desmoid tumors): an FNCLCC/French Sarcoma Group phase II trial with a long-term follow-up. Ann Oncol. 2011 Feb;22(2):452-7. doi: 10.1093/annonc/mdq341. Epub 2010 Jul 9. PMID 20622000
- [Result] Fayette J, Dufresne A, Penel N, et al.: Imatinib for the treatment of aggressive fibromatosis/desmoid tumors (AF/DT) failing local treatment: updated outcome and predictive factors for progression free survival: a FNCLCC French Sarcoma Group-GETO study. [Abstract] J Clin Oncol 25 (Suppl 18): A-10062, 560s, 2007.